CLINICAL TRIAL: NCT05471739
Title: Simultaneous Assessment of Coronary Microvascular Dysfunction and Ischemia With Non-obstructed Coronary Arteries With Intracoronary Electrocardiogram and Intracoronary Doppler
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Murat Sezer, MD, Professor, Istanbul University
Other Study IDs: 2019/1285
Record Dates: First submitted 2022-07-19; First posted 2022-07-25 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Coronary Microvascular Dysfunction; Coronary Microvascular Disease; Non-Obstructive Coronary Atherosclerosis; Microvascular Angina; Microvascular Coronary Artery Disease; Ischemic Heart Disease
Keywords: INOCA; ANOCA; CMD; Coronary Microvascular Dysfunction; Ischemia with non-obstructive coronary arteries; Coronary Microvascular Disease; Microvascular Angina
MeSH Terms: conditions — Microvascular Angina; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary Microvascular Dysfunction has been consistently shown to play a considerable role in pathophysiology of Ischaemia with non-obstructed coronary arteries (INOCA). While the both diagnoses are individually related to remarkably worse outcome, there is no available method to simultaneously determine INOCA-CMD endotypes in vessel level, during the invasive diagnosis.

The investigators hereby hypothesize that, combined intracoronary electrocardiogram (IC-ECG) (considering the high sensitivity and specificity of IC-ECG for studied vessel-territory) and intracoronary doppler can simultaneously and successfully identify vessel specific coronary microvascular dysfunction and resulting ischemia, which may potentially enable immediate diagnosis and endotyping of CMD-INOCA subgroups during the invasive assessment of first ANOCA episode, obviating the need for further ischemia-studies such es SPECT, which have considerably higher costs and lower sensitivity.

Major coronary arteries of patients aged between 18 - 75 without obstructing coronary artery disease who have previously documented ischemia with non-obstructed coronary arteries (INOCA) via coronary angiogram and myocardial perfusion scan will be evaluated simultaneously with IC-ECG and intracoronary Doppler during rest and under adenosine induced hyperaemia.

Performance of the combined system to identify Coronary Microvascular Dysfunction with structural and functional subgroups as defined by abnormal Coronary Flow Reserve (CFR) and Hyperemic Microvascular Resistance (HMR) and Ischemia in downstream territories of same vessel area (as defined by perfusion scan) is intended to be determined.

The investigators also intend to interrogate the possible relationship between dynamic changes in IC-ECG parameters and invasively obtained intracoronary hemodynamic data.

DETAILED DESCRIPTION:
Background and Rationale of Study

Coronary Microvascular Dysfunction has been consistently shown to play a considerable role in pathophysiology of Ischaemia with non-obstructed coronary arteries (INOCA). While the both diagnoses are individually related to remarkably worse outcome, there is no available method to simultaneously determine INOCA-CMD endotypes in vessel level, during the invasive diagnosis.

Hypothesis

The investigators hereby hypothesize that, combined intracoronary electrocardiogram (IC-ECG) (considering its high sensitivity for ischemia and specificity for studied vessel-territory) and intracoronary doppler can simultaneously and successfully identify vessel specific coronary microvascular dysfunction and resulting ischemia, which may potentially enable immediate diagnosis and endotyping of CMD-INOCA subgroups during the invasive assessment of first ANOCA episode, obviating the need for further ischemia-studies such as SPECT, which have considerably higher costs and lower sensitivity and requires more hospital visits.

Study Method

Major coronary arteries of patients aged between 18 - 75 without obstructing coronary artery disease who have previously documented ischaemia with non-obstructed coronary arteries (INOCA) via coronary angiogram and myocardial perfusion scan will be evaluated simultaneously with IC-ECG and intracoronary Doppler during rest and under adenosine induced hyperaemia after obtaining informed consent. Flow (APVr, APVh) data will be collected via intracoronary doppler during rest and adenosine induced hyperaemia in concordance with guidelines and Coronary Flow Reserve will be determined. Microvascular resistances (HMR, BMR) will be calculated with distal pressures and flow data.

Simultaneous with intracoronary Doppler, IC-ECG records will be obtained during rest and hyperaemia. Paper records will be digitized offline in MATLAB environment. Delta ST, Delta ST integral, Delta T, Delta T integral will be measured and calculated and quantified as continuous values.

All participants will be go through careful medical evaluation and presence of exclusion criteria will be assessed.

At the end of the data collection period, all available major coronary arteries are expected to have:

1. Myocardial Perfusion Scan result: whether they relate to (supply blood) ischemic territory.
2. Structural/Functional Microvascular Status: (CFR and HMR)

   -Definition of Coronary Microvascular Dysfunction and Subgroups: CMD is defined as CFR < 2.5. Those with concomitant HMR > 1.9 will be further labeled as structural CMD whereas vessels with CFR <2.5 and HMR <1.9 will be labeled as functional CMD.
3. IC-ECG parameters

ELIGIBILITY:
Inclusion Criteria:

* ≥1 previous episode of typical angina pectoris with normal coronary angiograms (Angina with Non-obstructed Coronary Arteries)
* positive myocardial perfusion scan (MPS) for ischemia or slow-flow.

Exclusion Criteria:

* obstructive epicardial coronary artery disease of at least 1 coronary artery in angiogram
* lung disease causing severe bronchospasm
* NYHA III - IV Heart Failure
* Bundle Branch Block
* Hb < 10 g/dL
* Active Malignancy
* Active Infection
* Morbid Obesity
* Pacemaker (Actively Pacing)
* Peripheral Artery Disease
* Previous CABG
* Chronic Hypoxia due to lung diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 - 75 years old patients with previously documented ischemia with non-obstructed coronary arteries and positive ischemia test (myocardial perfusion scan or slow-flow) to be enrolled. Patients meeting at least one exclusion criteria won't be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Hyperemic Microvascular Resistance (HMR) | Intraprocedural during coronary angiography
  the ratio of mean distal coronary pressure to average flow velocity
Coronary Flow Reserve (CFR) | Intraprocedural during coronary angiography
  the ratio between coronary blood flow at maximal hyperemia and at baseline condition
Delta ST | Intraprocedural during coronary angiography
  absolute shift of ST segment in IC-ECG record (at J point)
Delta ST Integral | Intraprocedural during coronary angiography
  absolute change in area between ST segment and isoelectric line

SECONDARY OUTCOMES:
Resting Average Peak Velocity | Intraprocedural during coronary angiography
Hyperemic Average Peak Velocity | Intraprocedural during coronary angiography

OTHER OUTCOMES:
Basal Microvascular Resistance (BMR) | Intraprocedural during coronary angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Jansen TPJ, Konst RE, Elias-Smale SE, van den Oord SC, Ong P, de Vos AMJ, van de Hoef TP, Paradies V, Smits PC, van Royen N, Damman P. Assessing Microvascular Dysfunction in Angina With Unobstructed Coronary Arteries: JACC Review Topic of the Week. J Am Coll Cardiol. 2021 Oct 5;78(14):1471-1479. doi: 10.1016/j.jacc.2021.08.028. PMID 34593129
- [Background] Ong P, Camici PG, Beltrame JF, Crea F, Shimokawa H, Sechtem U, Kaski JC, Bairey Merz CN; Coronary Vasomotion Disorders International Study Group (COVADIS). International standardization of diagnostic criteria for microvascular angina. Int J Cardiol. 2018 Jan 1;250:16-20. doi: 10.1016/j.ijcard.2017.08.068. Epub 2017 Sep 8. PMID 29031990
- [Background] Kunadian V, Chieffo A, Camici PG, Berry C, Escaned J, Maas AHEM, Prescott E, Karam N, Appelman Y, Fraccaro C, Louise Buchanan G, Manzo-Silberman S, Al-Lamee R, Regar E, Lansky A, Abbott JD, Badimon L, Duncker DJ, Mehran R, Capodanno D, Baumbach A. An EAPCI Expert Consensus Document on Ischaemia with Non-Obstructive Coronary Arteries in Collaboration with European Society of Cardiology Working Group on Coronary Pathophysiology & Microcirculation Endorsed by Coronary Vasomotor Disorders International Study Group. Eur Heart J. 2020 Oct 1;41(37):3504-3520. doi: 10.1093/eurheartj/ehaa503. PMID 32626906
- [Background] Bigler MR, Seiler C. Detection of myocardial ischemia by intracoronary ECG using convolutional neural networks. PLoS One. 2021 Jun 14;16(6):e0253200. doi: 10.1371/journal.pone.0253200. eCollection 2021. PMID 34125855
- [Derived] Cevik E, Tas A, Demirtakan ZG, Damman P, Alan Y, Broyd CJ, Ozcan A, Simsek DH, Sonsoz MR, Royen NV, Perera D, Davies JE, Umman S, Sezer M. Intracoronary electrocardiogram detects coronary microvascular dysfunction and ischemia in patients with no obstructive coronary arteries disease. Am Heart J. 2024 Apr;270:62-74. doi: 10.1016/j.ahj.2024.01.003. Epub 2024 Jan 25. PMID 38278503
- [Derived] Hasdemir H, Tas A, Cevik E, Alan Y, Broyd CJ, Ozcan A, Sonsoz MR, Kara I, Demirtakan ZG, Parker K, Perera D, Umman S, Sezer M. Primary versus iatrogenic (post-PCI) coronary microvascular dysfunction: a wire-based multimodal comparison. Open Heart. 2023 Nov 27;10(2):e002437. doi: 10.1136/openhrt-2023-002437. PMID 38011991